CLINICAL TRIAL: NCT06847035
Title: Efficacy Study of Oral Collagen Peptide on Skin Conditions
Brief Title: Efficacy Study of Oral Collagen Peptide on Skin Condition Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Meifute Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YKEC-2024-001
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Skin Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator (Active Comparator): collagen peptide solid beverage
  Interventions: Dietary Supplement: Active Comparator
- Placebo Comaprator (Placebo Comparator): placebo solid beverage
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Active Comparator — LISAVEI collagen peptide solid beverage ( contain 5 g collagen peptide)，once daily for 12 weeks
  Arms: Active Comparator
Dietary Supplement: Placebo Comparator — placebo solid beverage (Maltodextrin with edible flavor)，once daily for 12 weeks
  Other Names: placebo solid beverage
  Arms: Placebo Comaprator

SUMMARY:
To assess if oral intake of collagen peptide can improve skin conditions such as skin thickness, density and firmness.

DETAILED DESCRIPTION:
This is an one site, randomized, double-blind controlled clinical trial to assess the oral supplement of LISAVEI collagen peptide solid beverage on skin ageing improvement. Study product with collagen peptide and placebo product without collagen were randomly assigned to 90 eligible participants enrolled according to the inclusion and exclusion criteria. They took the assigned product once daily dissolved in 100 ml warm water for 12 weeks with 4-week regression phase(without intake of the test products), and visit the study site in Shanghai for four times(before starting the treatment, after 8 and 12 weeks, and 4 weeks after the last intake). Skin measurements including skin firmness, skin density, skin hydration and skin barrier were carried out at each visit with professional equipment and imaging system. Data were analyzed to validate if the administration of the test collagen peptide solid beverage will improve skin aging parameters such as firmness, thickness, density, hydration and skin barrier compared to placebo. The lasting effect was also observed by comparing between the two groups after 4-week regression time.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female adults aged between 35-55 years old
2. With fine wrinkles and skin laxity
3. Personal informed consents to participate in the study
4. Agree to keep their daily skincare routine unchanged for the duration of the study
5. Maintain good sun protection habits

5. Agree to refrain from wearing make-up on the face on the each study visit

Exclusion Criteria

1. Female who is pregnant or nursing or planning to become pregnant during the course of the study
2. Individuals who are in the perimenopausal stage.
3. BMI<18.5 or BMI >27.9
4. Individuals suffering from chronic systemic diseases such as cardiovascular, cerebrovascular, liver, and kidney diseases.
5. Individuals who have diabetes.
6. Individuals suffering from skin conditions such as psoriasis, eczema, atopic dermatitis, and severe acne.
7. Individuals with depression or sleep disorders, those who smoke, and those who abuse alcohol.
8. Individuals who are using hormonal drugs, medications for obesity, absorption inhibitors, antidepressants, or appetite suppressants.
9. Individuals who have used hormones or anti-inflammatory drugs on their face and upper arms within the past two months.
10. Individuals who received facial laser therapy, chemical peeling or UV overexposure in the past 3 months
11. Individuals who can not avoid prolonged exposure to sunlight.
12. Individuals who are currently participating in other clinical studies or trials.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Skin firmness | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  The changes of skin firmness parameter tested by Cutometer MPA580
Skin thickness | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  The changes of skin thickness （μm） tested by Ultrascan UC 22
Skin density | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  The changes of skin density tested by Ultrascan UC 22

SECONDARY OUTCOMES:
Skin hydration | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  The changes of skin hydration tested by Corneometer CM825
Skin barrier | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  The changes of Trans Epidermal Water Loss (skin barrier parameter) tested by Tewameter TM300
Facial image | before product treatment (T 0), after 8 weeks(T 1)and 12 weeks(T 2) of daily product intake, 4 weeks after the last intake(T 3, 4-week regression phase)
  Photo documents of left, right and frontal facial views

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fumei Dermatology Clinic, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang Y, Zhu W, Luo W, Ma Y, Zhou Y. The Sustained Effects of Bioactive Collagen Peptides on Skin Health: A Randomized, Double-Blind, Placebo-Controlled Clinical Study. J Cosmet Dermatol. 2025 Dec;24(12):e70565. doi: 10.1111/jocd.70565. PMID 41311286